CLINICAL TRIAL: NCT02599636
Title: Multicenter Prospective Study: To Survive After ICU Discharge
Brief Title: To Survive After ICU Discharge
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Althaia Xarxa Assistencial Universitària de Manresa (Other)
Responsible Party: Principal Investigator, Silvia Cano Hernández, Physician, Althaia Xarxa Assistencial Universitària de Manresa
Other Study IDs: Althaia
Record Dates: First submitted 2015-10-30; First posted 2015-11-06 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: In-Hospital Mortality; Number of ICU Readmission; Number of Warnings On-duty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: None intervention — Investigators will study the usual medical assistance

SUMMARY:
Many factors before and after ICU stay determine the outcome of patients at ICU discharge, the type of illness, physical dependence and other sequelae can be a trigger for complications in hospital ward which can induce ICU readmission and worse outcome. The quality of medical assistance during all the hospitalisation should be guaranteed and many complications or fatal events could be avoidable.

The objective of the present study is to demonstrate that collaboration between the intensivist and other medical teams in ward can reduce ICU readmission and hospital mortality after ICU discharge.

DETAILED DESCRIPTION:
Material and Methods This observational multicenter study will be done in 21 medical-surgical ICUs. We will use Sabadell Score like prognostic scale at ICU discharge and the intensivist will collaborate with the medical team in medical assistance of patients at risk (Sabadell Score 1 and 2). Investigators will compare the hospital mortality and the readmission rate with a previous period when this collaboration didn't exist.

Anticipate results The collaboration of attending intensivist might reduce ward mortality after ICU discharge by 3%.

ELIGIBILITY:
Inclusion Criteria:

* All patients with Sabadell Score 1 (poor prognosis in long term) and 2 (poor prognosis in short term) at ICU discharge

Exclusion Criteria:

* patients younger than 18 years old
* patients with Sabadell Score 0 (good prognosis)
* patients with Sabadell Score 3 (null expected survival)
* patients transferred to other hospitals

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients at ICU discharge
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The decline in hospital mortality | 3 months

SECONDARY OUTCOMES:
The decline in number of warnings on-duty | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Cano Hernández, Physician, Principal Investigator — Althaia Xarxa Assistencial Universitaria de Manresa
Locations (1):
- Althaia Xarxa Assistencial Universitaria de Manresa, Manresa, Barcelona, Spain